CLINICAL TRIAL: NCT06161961
Title: Interventional Pilot Study on the Evaluation of Functionality, Degree of Safety and Reliability of a New Robotic Prosthesis for Treatment of Transtibial Lower Limb Amputations
Brief Title: Interventional Study on the Evaluation of Functionality, Safety of a Robotic Prosthesis for Transtibial Amputations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Claudio Macchi, Full Professor, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MOTU TT - studio clinico
Record Dates: First submitted 2023-11-08; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Amputation; Amputation; Traumatic, Leg, Lower
Keywords: lower limb; transtibial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prosthetic group (Experimental): prosthetic group performs the entire protocol with the prosthesis prototype.
  Interventions: Device: WRL TTP

INTERVENTIONS:
Device: WRL TTP — evaluation of functionality, degree of safety and reliability of the lower limb prosthesis prototype

SUMMARY:
The goal of this multicenter interventional pilot is to verify the functionality of a prosthesis for trans-tibial amputees.

The main question it aims to answer are:

* Is to verify the technical functionality, safety and reliability of the propulsive lower limb prosthesis prototype, with active ankle, so as to provide indications regarding the technical and functional developments to be implemented in the finalization of the device.
* Provide an indication of the functional effectiveness of the device and its satisfaction by patients.

Participants will perform:

* walking tests inside parallel bars on flat and/or inclined terrain;
* walking tests on treadmill;
* stair climbing/descent tests.

ELIGIBILITY:
Inclusion Criteria:

* Trans-tibial lower limb amputation;
* Medicare functional classification: Level K3-K4;
* Subjects who have worn prostheses for at least 1 year (experienced wearers);
* Use of prosthesis with energy-returning prosthetic foot.

Exclusion Criteria:

* Relevant medical comorbidities (serious neurological pathologies, cardiovascular pathologies, diabetes/hypertension not stabilized, severe sensory deficits);
* Wearers of implantable cardiac medical devices (PMK or AICD);
* Cognitive impairment (MMSE corrected for age and education <24);
* Inability or unavailability to provide informed consent;
* Severe depressive and/or anxious symptoms.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
ad hoc check-list Adverse Event | baseline
  questionnaire that evaluate the device feasability of the prosthesis and description of any adverse events.
ad hoc check-list Adverse Event | day 2
  questionnaire that evaluate the device feasability of the prosthesis and description of any adverse events.
ad hoc check-list Adverse Event | day 3
  questionnaire that evaluate the device feasability of the prosthesis and description of any adverse events.
ad hoc check-list Adverse Event | day 4
  questionnaire that evaluate the device feasability of the prosthesis and description of any adverse events.
ad hoc check-list Adverse Event | day 5
  questionnaire that evaluate the device feasability of the prosthesis and description of any adverse events.

SECONDARY OUTCOMES:
CR-10 Borg Scale | day 5
  0-10 numerical rating scale that evaluate of the subjective perception of effort during walking
System usability scale | baseline
  a questionnaire made up of 10 questions whose answers are yes structured on a Likert scale with values 0-100 that assess the usability of the prosthesis
System usability scale | day 5
  a questionnaire made up of 10 questions whose answers are yes structured on a Likert scale with values 0-100 that assess the usability of the prosthesis
10mwt - 10 meters walking test | day 2
  to assess the walking speed
10mwt - 10 meters walking test | day 3
  to assess the walking speed
SCT - stair climb test | day 2
  to assess the capability of climb 8 stairs
SCT - stair climb test | day 3
  to assess the capability of climb 8 stairs
TUG - Timed Up and GO | day 2
  to assess lower limb capability
TUG - Timed Up and GO | day 3
  to assess lower limb capability
6mwt - 6 minute walking test on the treadmill | day 4
  to assess the fatigue
6mwt - 6 minute walking test on the treadmill | day 5
  to assess the fatigue
Gait analisys | day 5
  to assess the gait pattern

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Au SK, Herr H, Weber J, Martinez-Villalpando EC. Powered ankle-foot prosthesis for the improvement of amputee ambulation. Annu Int Conf IEEE Eng Med Biol Soc. 2007;2007:3020-6. doi: 10.1109/IEMBS.2007.4352965. PMID 18002631
- [Background] Buckley JG, O'Driscoll D, Bennett SJ. Postural sway and active balance performance in highly active lower-limb amputees. Am J Phys Med Rehabil. 2002 Jan;81(1):13-20. doi: 10.1097/00002060-200201000-00004. PMID 11807327
- [Background] Borg, G. (1998). Borg's Perceived Exertion and Pain Scales. Human Kinetics.
- [Background] Brooke, J. (1996). SUS: a
- [Background] Cherelle P, Grosu V, Matthys A, Vanderborght B, Lefeber D. Design and Validation of the Ankle Mimicking Prosthetic (AMP-) Foot 2.0. IEEE Trans Neural Syst Rehabil Eng. 2014 Jan;22(1):138-48. doi: 10.1109/TNSRE.2013.2282416. Epub 2013 Oct 7. PMID 24122571
- [Background] Eslamy, M., Grimmer, M., & Seyfarth, A. (2012). Effects of Unidirectional Parallel Springs on Required Peak Power and Energy in Powered Prosthetic Ankles: Comparison between Different Active Actuation Concepts. Proceedings of the 2012 IEEE International Conference on Robotics and Biomimetics, December 11-14, Guangzhou, China.
- [Background] Gailey R, Allen K, Castles J, Kucharik J, Roeder M. Review of secondary physical conditions associated with lower-limb amputation and long-term prosthesis use. J Rehabil Res Dev. 2008;45(1):15-29. doi: 10.1682/jrrd.2006.11.0147. PMID 18566923
- [Background] Grimmer, M., & Seyfarth, A. (2014). Mimicking human-like leg function in prosthetic limbs. In Neurorobotics: from brain machine interfaces to rehabilitation robotics. Berlin: Springer.
- [Background] Grimmer, M., Eslamy, M., & Seyfarth, A. (2014). Energetic and Peak Power Advantages of Series Elastic Actuators in an Actuated Prosthetic Leg for Walking and Running. Actuators, 3:1-19.
- [Background] Huang S, Huang H. Voluntary Control of Residual Antagonistic Muscles in Transtibial Amputees: Reciprocal Activation, Coactivation, and Implications for Direct Neural Control of Powered Lower Limb Prostheses. IEEE Trans Neural Syst Rehabil Eng. 2019 Jan;27(1):85-95. doi: 10.1109/TNSRE.2018.2885641. Epub 2018 Dec 7. PMID 30530332
- [Background] Mak AF, Zhang M, Boone DA. State-of-the-art research in lower-limb prosthetic biomechanics-socket interface: a review. J Rehabil Res Dev. 2001 Mar-Apr;38(2):161-74. PMID 11392649
- [Background] Marino, M., Pattni, S., Greenberg, M., Miller, A., Hocker, E., Ritter, S., et al. (2015). Access to prosthetic devices in developing countries: Pathways and challenges. 2015 IEEE Global Humanitarian Technology Conference (GHTC), 45-51.
- [Background] Pirouzi G, Abu Osman NA, Eshraghi A, Ali S, Gholizadeh H, Wan Abas WA. Review of the socket design and interface pressure measurement for transtibial prosthesis. ScientificWorldJournal. 2014;2014:849073. doi: 10.1155/2014/849073. Epub 2014 Aug 13. PMID 25197716
- [Background] Segal AD, Orendurff MS, Klute GK, McDowell ML, Pecoraro JA, Shofer J, Czerniecki JM. Kinematic and kinetic comparisons of transfemoral amputee gait using C-Leg and Mauch SNS prosthetic knees. J Rehabil Res Dev. 2006 Nov-Dec;43(7):857-70. doi: 10.1682/jrrd.2005.09.0147. PMID 17436172